CLINICAL TRIAL: NCT00551291
Title: An Open Label Study of the Effects of a Combination of NeoRecormon, CellCept and Prednisone on Hematological Parameters and Cytogenesis in Patients With Low or Intermediate Risk Myelodysplastic Syndromes.¿
Brief Title: A Study of NeoRecormon (Epoetin Beta), CellCept (Mycophenolate Mofetil) and Prednisone in Patients With Low or Intermediate Myelodysplastic Syndromes.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20559
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Mycophenolic Acid; Prednisone; epoetin beta

ARMS (1):
- Mycophenolate Mofetil + Prednisone + Erythropoietin Beta (Experimental): Mycophenolate mofetil (MMF) 1 gm twice daily orally and prednisone 10 mg/day orally until the end of the study. Recombinant human erythropoietin beta 30,000 IU/week, subcutaneously for 6 weeks was added in case of no significant response at Week 12.
  Interventions: Drug: Mycophenolate mofetil; Drug: Prednisone; Drug: Erythropoietin Beta

INTERVENTIONS:
Drug: Mycophenolate mofetil — 1 gm twice daily orally until end of study.
  Other Names: CellCept; MMF
Drug: Prednisone — 10 mg/day orally until end of study.
Drug: Erythropoietin Beta — Recombinant human erythropoietin beta at doses of 30,000 IU/week by the subcutaneous route for 6 weeks.
  Other Names: NeoRecormon

SUMMARY:
This single arm study will evaluate the efficacy and safety of a combination of NeoRecormon, CellCept and prednisone in patients with low or moderate risk myelodysplastic syndromes (MDS). In the first phase of the study, patients will receive CellCept (1g p.o. twice daily) plus prednisone. After 3 months, if patients have not responded to treatment, NeoRecormon (30000 IU/week, s.c.) will be added to the treatment regimen. If there is no response to NeoRecormon after 6 weeks, the dose will be increased to 60000 IU/week. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* diagnosis of MDS, according to International Prognostic Scoring System (IPSS) criteria;
* low or intermediate risk, who are not candidates for treatment with growth factors, or who have not responded to these treatments.

Exclusion Criteria:

* previous treatment with CellCept, or any erythropoietin-stimulating drug;
* diagnosis of proliferative chronic myelomonocytic leukemia;
* prior or concomitant malignancies other than MDS, with the exception of basocellular, spinocellular or adequately treated in situ cervical cancer, in the past 3 years;
* biological antitumor and myelosuppressive treatment within 28 days before start of study;
* bone marrow precursor cell transplantation previous to study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Spain (5):
  - Barakaldo
  - Barcelona
  - Cadiz
  - Madrid
  - Palma de Mallorca

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mycophenolate Mofetil + Prednisone + Erythropoietin Beta
Started | 10
Completed | 9
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mycophenolate Mofetil + Prednisone + Erythropoietin Beta
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.00 (5.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Response as Measured by the International Working Group (IWG) Criteria for Hematological Improvement
Description: International Working Group (IWG) criteria for hematological improvement was defined as having hemoglobin (Hgb) <11 g/dL (pretreatment) and an increase in Hgb ≥1.5 g/dL after ≥8 weeks of treatment.
Time Frame: Up to approximately 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Mycophenolate Mofetil + Prednisone + Erythropoietin Beta
Number analyzed (Participants) | 10
percentage of participants
  Week 12 (n=4) | 50.00
  Week 18 (n=7) | 71.43
  End of study (n=3) | 100.00

2. Primary Outcome: Mean Number of Blood Transfusions Per Visit
Time Frame: Up to approximately 2 years
Measure: Mean (Standard Deviation); unit: transfusions/visit
Arm/Group | Mycophenolate Mofetil + Prednisone + Erythropoietin Beta
Number analyzed (Participants) | 10
transfusions/visit
  Baseline (n=8) | 4.13 (2.30)
  Week 12 (n=6) | 5.83 (2.86)
  Week 18 (n=5) | 2.80 (1.92)
  End of Study (n=3) | 2.33 (1.53)

3. Secondary Outcome: Percentage of Participants With at Least One Adverse Event (AE)
Description: An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study and laboratory or clinical tests that resulted in a change in treatment or discontinuation from study drug were reported as adverse events.
Time Frame: Up to approximately 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Mycophenolate Mofetil + Prednisone + Erythropoietin Beta
Number analyzed (Participants) | 10
percentage of participants | 90.00

ADVERSE EVENTS:
Time Frame: Up to approximately 2 years.
Arm/Group | Mycophenolate Mofetil + Prednisone + Erythropoietin Beta
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mycophenolate Mofetil + Prednisone + Erythropoietin Beta (N=10)
Pneumonia (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Cardiac insufficiency (Cardiac disorders) | 1
Colecistitis (Hepatobiliary disorders) | 1
Achilles tendon´s break (Musculoskeletal and connective tissue disorders) | 1
Rectal bleeding (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mycophenolate Mofetil + Prednisone + Erythropoietin Beta (N=10)
Upper respiratory tract catarrh (Infections and infestations) | 3
Respiratory infection (Infections and infestations) | 1
Bronchial infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Herpes labialis (Infections and infestations) | 1
Diarrhea (Gastrointestinal disorders) | 2
Gastroenteritis (Gastrointestinal disorders) | 1
Epigastralgia (Gastrointestinal disorders) | 1
Dyspnea on exertion (Cardiac disorders) | 1
Dyspnea to great efforts (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Achilles tendon´s tendinitis (Musculoskeletal and connective tissue disorders) | 1
Coxalgia (Musculoskeletal and connective tissue disorders) | 1
Asthenia (General disorders) | 2
Dysthermia feeling (General disorders) | 1
Facial allergic reaction (Skin and subcutaneous tissue disorders) | 1
Occasional tightness in the chest (Respiratory, thoracic and mediastinal disorders) | 1
Nervousness (Psychiatric disorders) | 1
Chest injury due to fall (Injury, poisoning and procedural complications) | 1
Decompensated diabetes mellitus (Endocrine disorders) | 1
Splenomegaly increase (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.